CLINICAL TRIAL: NCT03143348
Title: Prognostic Markers of Inflammation in Infants Undergoing Cardiopulmonary Bypass (ProCard): an Observational Pilot Study
Brief Title: Prognostic Markers of Inflammation in Infants Undergoing Cardiopulmonary Bypass
Acronym: ProCard
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 7676
Record Dates: First submitted 2017-03-13; First posted 2017-05-08 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Congenital Heart Defect; Cardiopulmonary Bypass; Inflammatory Response; Low Cardiac Output Syndrome; Inflammation
MeSH Terms: conditions — Heart Defects, Congenital; Cardiac Output, Low; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control/Nonsurgical: Infants with postnatally confirmed acyanotic congenital heart disease not expected to require surgery in the first six months of life.
  Interventions: Procedure: Single blood draw
- Surgery w/o bypass: Infants with postnatally confirmed congenital heart disease requiring cardiac surgery without cardiopulmonary bypass.
  Interventions: Procedure: Multiple blood draws
- Surgery w/ bypass: Infants with postnatally confirmed congenital heart disease requiring cardiac surgery with cardiopulmonary bypass.
  Interventions: Procedure: Multiple blood draws

INTERVENTIONS:
Procedure: Single blood draw — One blood draw of 0.5 ml volume prior to discharge
  Groups: Control/Nonsurgical
Procedure: Multiple blood draws — Blood draw at 6 peri-operative time points.
  Groups: Surgery w/o bypass
Procedure: Multiple blood draws — Blood draw at 7 peri-operative time points
  Groups: Surgery w/ bypass

SUMMARY:
This study evaluates the effect of heart-lung bypass on babies undergoing cardiac surgery. The investigators want to learn more about the inflammation that exposure to bypass creates in the body by studying markers of inflammation and cell injury in the bloodstream. Additionally, the investigators want to examine if these markers can predict which babies develop post-surgical complications. The hypothesis is that babies who undergo bypass will have higher levels of these markers than babies not exposed to bypass and that these markers will correlate with how the baby does clinically after surgery.

This study will evaluate markers via blood sampling in babies with congenital heart disease who do not undergo cardiac surgery, those that undergo surgery without bypass, and those that undergo surgery with bypass. The overall goal is that this study will lead to useful biomarkers and lay the groundwork for future novel therapies aimed at improving outcomes for babies who require heart-lung bypass.

DETAILED DESCRIPTION:
This is a minimal risk observational study looking at markers of inflammation and cell injury in the bloodstream of babies with congenital heart disease, with a particular emphasis on whether these markers can predict low cardiac output syndrome in infants who undergo heart-lung bypass. Low cardiac output syndrome is a common postoperative complication marked by poor blood flow to the body affecting nearly 1/3 of infants post-bypass and is associated with significant morbidity and mortality.

Babies not requiring surgery will serve as the control group. Infants in group 1 will have 0.5 ml of blood drawn prior to discharge. This will be scavenged from the laboratory when possible. Infants in groups 2 and 3 will require serial blood draws over peri-operative time points each in the volume of 0.5 ml.

Group 2:

T0 = Before surgery (in the OR) T1 = After chest closure or end of case (in the OR) T2 = On admission to the pediatric intensive care unit T3 = Timed 4-6 hours after the time of admission T4 = Timed 12 hours (+/- 1 hour) after the time of admission T5 = Timed 24 hours (+/-1 hour) after the time of admission

Group 3:

T0 =Pre-cardiopulmonary bypass to be obtained in the operating room just prior to surgery T1 = After going on bypass (but prior to modified ultrafiltration) T2 = After modified ultrafiltration T3 = On admission to the pediatric intensive care unit T4 = Timed 4-6 hours after the time of admission T5 = Timed 12 hours (+/- 1 hour) after the time of admission T6 = Timed 24 hours (+/-1 hour) after the time of admission

ELIGIBILITY:
Inclusion Criteria:

* Infants < 6 months of age
* Born at ≥ 36 weeks gestational age
* Birth weight ≥ 2.5 kilograms
* Postnatally confirmed congenital heart disease by echocardiogram

Exclusion Criteria:

* Requiring ≥ 2 vasopressors prior to surgery
* Preoperative proven sepsis within one week of surgery
* Prior surgery within one week of cardiac repair (except PA banding which is not excluded)
* Cardiac catheterization within one week of surgery
* Significant extra-cardiac anomalies that may impair organ function

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants <6 months of age with congenital heart disease at OU Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-06-04 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Biomarker levels and their relationship to LCOS | Baseline level and described time points over the first twenty-four hours postoperatively
  Changes in markers of inflammation and cell injury (histones, IL-6, etc.) and correlation with patients who develop low cardiac output syndrome

SECONDARY OUTCOMES:
Change in level of inflammatory response | Baseline, up to 24 hours
  Changes in markers of inflammation and cell injury (IL-6, IL-8, etc.) in the peri-operative period (prior to surgery up to 24 hours postop)
Length of mechanical ventilation | Participants will be followed throughout hospital course, maximum length of follow-up one year
  Number of days on mechanical ventilation following day of surgery until the point of extubation
Acute kidney injury | Participants will be followed for the first twenty four hours postoperatively
  Doubling of creatinine in first twenty four hours compared to preoperative levels
Extracorporeal membrane oxygenation (ECMO) | First 48 hours postoperatively
  Whether or not patient requires ECMO cannulation
ICU length of stay | Participants will be followed throughout PICU/CVICU stay, maximum length of follow-up one year
  Number of days requiring pediatric/cardiac intensive care unit following day of surgery
Hospital length of stay | Participants will be followed throughout entire hospital course, maximum length of follow-up one year
  Number of hospital days patient requires following the day of surgery
Mortality risk | PIM-2 calculated within one hour of admission to PICU and PRISM-3 calculated at 12 and 24 hours after PICU admission
  Pediatric risk of mortality-3 scale (PRISM-3) and pediatric index of mortality (PIM-2)
Mortality | Participants will be followed throughout hospital course, maximum length of follow-up one year
  Any type of death that occurs during patient's hospitalization
Low cardiac output syndrome | Assessed at 48 hours postoperatively
  At least two of the following criteria at any post-operative time point within the first twenty four hours: (a) prolonged cap refill >3 sec, SBP <5th %ile for age and gender, low UOP <1 cc/kg/hr for at least 6 hr not responsive to diuretics, persistently elevated arterial lactate >2 and metabolic acidosis defined as an increase in the base deficit of >4, inotropic score >20, cardiac arrest within 48 hr after surgery, or the need for extracorporeal membrane oxygenation (ECMO) for hemodynamic instability within 48 hours postop

CONTACTS AND LOCATIONS:
Overall Officials: Hala Chaaban, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No